CLINICAL TRIAL: NCT05771025
Title: Effect of Hepatectomy on the Prognosis of Patients With Nasopharyngeal Carcinoma Liver Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWK-2022-7275
Record Dates: First submitted 2023-02-06; First posted 2023-03-16 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Nasopharyngeal Carcinoma; Liver Metastases
Keywords: Nasopharyngeal Carcinoma; Liver Metastases; Hepatectomy; Prognosis
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatectomy group (Experimental): Patients in the hepatectomy group receive hepatectomy, which could be combined with radiotherapy and chemotherapy for the primary tumor during the perioperative period.
  Interventions: Procedure: Hepatectomy

INTERVENTIONS:
Procedure: Hepatectomy — Patients in the hepatectomy group receive liver resection.

SUMMARY:
The goal of this clinical trial is to learn about hepatectomy on the prognosis of patients with nasopharyngeal carcinoma liver metastases (NCLM). The main questions it aims to answer are:

To explore the effect of hepatectomy on the overall survival, recurrence-free survival and other prognostic indicators of patients with NCLM.

To explore the impact of hepatectomy on the safety of patients with NCLM.

Researchers will compare the prognosis of the patients in the hepatectomy group and the patients with NCLM who were prospectively enrolled in the same institution and received only systemic treatment at the same time by propensity score matching.

ELIGIBILITY:
Inclusion Criteria:

* Nasopharyngeal carcinoma liver metastases (NCLM) are diagnosed by pathological confirmation of liver biopsy or imaging findings combined with clinical history.
* ECOG score ≤ 2 points.
* 1. Patients with no recurrence of the primary tumor and oligometastasis in the liver. 2. Patients with multiple metastases (bone) without primary tumor recurrence and liver metastases have stable disease (SD) or partial remission (PR) or complete remission (CR) after systemic treatment except for liver lesions. 3. Patients with primary tumor recurrence and liver metastasis (may be combined with bone metastasis) have SD or PR or CR after systemic treatment except for liver lesions.
* Able to perform radical resection of liver lesions.
* Good liver function (Child-Pugh grade A liver function, estimated remaining liver volume ≥ 30%).
* Blood test, coagulation function, liver and kidney function, electrocardiogram, chest X-ray and other preoperative examinations show no clear contraindications for surgery.
* Expected survival ≥ 6 months.
* Those who voluntarily participate in this study and signe the informed consent form.

Exclusion Criteria:

* Younger than 18 or older than 70 years old.
* ECOG score > 2 points.
* Combined with distant metastasis other than liver and bone.
* Disease progression (PD) after systemic treatment of the primary tumor and bone metastases.
* The liver lesion cannot be resected by R0.
* Insufficient liver reserve function (preoperative liver function Child-Pugh B or C grade and cannot be reduced to A grade in a short time, or estimated remaining liver volume <30%).
* Combined with surgical contraindications in the preoperative examination, such as cardiac clinical symptoms or diseases that are not well controlled, abnormal coagulation function with bleeding tendency, or receiving thrombolytic therapy, etc..
* Liver metastases have received local treatment for liver metastases such as interventional and radiofrequency.
* Pregnant or lactating women.
* History of malignant tumors in other parts, severe mental illness, etc..
* Patients or family members cannot understand the conditions and objectives of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival time | up to 60 months
  Refers to the time from liver resection to death from any cause.

SECONDARY OUTCOMES:
Intrahepatic recurrence-free survival | up to 60 months
  Refers to the time from the start of liver resection to the date of confirmation of intrahepatic tumor recurrence or death from any cause, whichever is earlier, in patients who underwent hepatectomy.
Perioperative morbidity rate | 3 months
  Refers to the incidence of perioperative complications.
Perioperative mortality rate | 1 month
  Refers to the mortality rate of patients within 30 days after liver resection.
Unplanned reoperation rate | 1 month
  Refers to the unplanned reoperation rate due to various reasons during the same hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Wang, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
We can share IPD with other researchers under reasonable requests.